CLINICAL TRIAL: NCT05793658
Title: Is Respiratory Rate Derived From Capnography Can Prevent Adverse Events Occurred in Sedated Patients.
Brief Title: Role of Respiratory Rate Derived From Capnography in Sedated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al Jedaani Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1/5/22
Record Dates: First submitted 2023-02-28; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Sedation Problems
Keywords: Sedation; capnography; Respiratory rate; colonoscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedation with standard capnography (Active Comparator): 37 patient Sedation using midazolam + propofol for colonoscopy
  Interventions: Procedure: Standard capnography
- Sedation with modified capnography (Active Comparator): 37 patients in Sedation using midazolam + fentanyl + propofol for colonoscopy
  Interventions: Procedure: Modified capnography

INTERVENTIONS:
Procedure: Standard capnography — Patients undergoing colonoscopy under sedation were randomly assigned to receive standard capnography monitoring or modified capnography monitoring which can be achieved by tucking capnography probe under the face mask.74 patients were enrolled. Patient characteristics were well balanced between the two groups 37 patients in each group.
  Other Names: Qualitative capnograpyhy
  Arms: Sedation with standard capnography
Procedure: Modified capnography — If Respiratory rate below 14 b/m: more sedation isn't not advised and the patient may develop airway obstruction and needs airway intervention ( like jaw thrust or oral airway) If respiratory rate more than 20 b/m it means this patient is prone to awake or to move and this patient in need for incremental dose of sedative drug ( e.g 20 to 30 mg propofol) Also roughly speaking respiratory rate from 16 to 18 b/m is the target
  Other Names: Quantitative capnography
  Arms: Sedation with modified capnography

SUMMARY:
Although appropriate sedation is recommended during colonoscopy, patients are at risk for adverse events e.g hypoventilation and hypoxemia due to inadvertent oversedation. The aim of this study was to evaluate the benefit of additional quantitative capnography monitoring ( respiratory rate )in management of patient undergoing colonoscopy under sedation in preventing or reducing the incidence of adverse events and also determine when to start the procedure and when to give and not to give increments of sedative drugs during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 and 2 adult patients
* Age from 20 to 50 years old
* elective colonoscopy

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) above Class II
* History of psychiatric or neurological disease

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Hypoxemia | 1 hours
  Detected by pulse oximeter

SECONDARY OUTCOMES:
Patient movements during the procedure | 1 hour
  Measured by questionnaire to the gastroenterologist (scale from 1 to 5)
Effort exerted by the anesthesiologist ( the provider) | 1 hour
  Measured by questionnaire ( scale from 1 to 5 )
Patient satisfaction | 1 hour
  Measured by questionnaire ( scale from 1 to 5 )
Gastroenterologist satisfaction | 1 hour
  Measured by questionnaire ( scale from 1 to 5 )

CONTACTS AND LOCATIONS:
Locations (1):
- Al Jedaani group of hospitals, Jeddah, Meccah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No